CLINICAL TRIAL: NCT04597476
Title: A Randomized, Double-blind Study to Evaluate the Clinical Effect and Safety of Fucoidan in Patients With Squamous Cell Carcinomas of the Head and Neck
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hi-Q Marine Biotech International, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HIQ-FUCO-02
Record Dates: First submitted 2020-09-29; First posted 2020-10-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Squamous Cell Carcinomas of the Head and Neck
MeSH Terms: interventions — fucoidan

STUDY DESIGN:
Intervention Model Description: Fucoidan Group: Fucoidan 4.4 g, PO, bid for 24 weeks Placebo Group: Potato starch 4.4 g, PO, bid for 24 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be centrally randomized in a 1:1 ratio to receive either Fucoidan or placebo (potato starch) Eligible subjects will receive fucoidan twice daily (BID) in combination with chemotherapy and radiation therapy over a 24-week treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fucoidan Group (Experimental): Fucoidan powder at 4.4 g per sachet (dose) for oral administration. Fucoidan 4.4 g, PO, bid for 24 weeks
  Interventions: Dietary Supplement: Fucoidan
- Potato starch (Placebo Comparator): Potato starch at 4.4 g per sachet (dose) for oral administration. Potato starch 4.4 g, PO, bid for 24 weeks
  Interventions: Other: Placebo( Potato starch)

INTERVENTIONS:
Dietary Supplement: Fucoidan — Fucoidan refers to a class of fucose-enriched sulfated polysaccharides with an average molecular weight of 20,000 Daltons (Da), which can be found in many varieties of edible brown seaweeds and algae . In cell culture studies and animal studies, fucoidan has been shown to possess a range of biological activities, including anti-cancer, anti-inflammatory, and immunoregulatory effects . A recent in vitro study conducted in head and neck squamous cell carcinoma (HNSCC) cell lines (H103, FaDu, and KB) showed that fucoidan could induce cell cycle arrest and possibly apoptosis in a dose-dependent manner, while also enhancing response to cisplatin treatment . In addition, fucoidan has also been shown to inhibit the proliferation of nasopharyngeal carcinoma cells and MC3 human mucoepidermoid carcinoma (MEC) cells .
  Arms: Fucoidan Group
Other: Placebo( Potato starch) — Potato starch 4.4gram
  Arms: Potato starch

SUMMARY:
This phase II study is a randomized, double-blind study that seeks to evaluate the clinical effects and safety of fucoidan in the treatment of cancer patients with stage III/IV head and neck squamous cell carcinoma.

Patients will be centrally randomized in a 1:1 ratio to receive either Fucoidan or placebo (potato starch) Eligible subjects will receive fucoidan twice daily (BID) in combination with chemotherapy and radiation therapy over a 24-week treatment period.

Clinical effects and safety parameters for all subjects who complete the treatment period will be followed for an additional 72 weeks after the treatment period.

DETAILED DESCRIPTION:
This phase II study is a randomized, double-blind study that seeks to evaluate the clinical effects and safety of fucoidan in the treatment of cancer patients with stage III/IV head and neck squamous cell carcinoma.

Patients will be centrally randomized in a 1:1 ratio to receive either Fucoidan or placebo (potato starch) Eligible subjects will receive fucoidan twice daily (BID) in combination with chemotherapy and radiation therapy over a 24-week treatment period.

Clinical effects and safety parameters for all subjects who complete the treatment period will be followed for an additional 72 weeks after the treatment period.

The total length of the study for each subject will be approximately 100 weeks, comprising the following time periods: screening period (28 days), treatment period (24 weeks), and follow-up period (72 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. The patients with stage III/IV head and neck squamous cell carcinoma (HNSCC) withoutdistant metastasis who had not received any treatment to head and neck cancer can be enrolled in this study.
2. Completed a computed tomography (CT) or magnetic resonance imaging (MRI) scan of the head and neck (including the primary tumor and neck nodes) within 6 weeks prior to enrollment.
3. Adequate renal function, with serum creatinine ≤ 1.5 mg/dL. Patients with serum creatinine > 1.5 mg/dL may be eligible if calculated creatinine clearance ≥ 55 mL/min as based on the results of the Cockcroft-Gault Equation or 24-hour urine collection.
4. Age ≥ 20 years and ≤ 75 years.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status = 0-1.
6. Expected lifespan > 6 months.
7. Adequate bone marrow function, as defined by absolute neutrophil count ≥ 1,500/μL, platelet count ≥ 100,000/μL, and hemoglobin ≥ 9 g/dL.
8. Adequate hepatic function, with total bilirubin ≤ 1.5 × upper normal limit (UNL; patients with hyperbilirubinemia caused by Gilbert's syndrome may be eligible if total bilirubin ≤ 2.5 × UNL), aspartate aminotransferase (AST) ≤ 2.5 × UNL, alanine aminotransferase (ALT) ≤ 2.5 × UNL, and alkaline phosphatase (ALP) ≤ 2.5 × UNL.
9. Men and women of childbearing potential must consent to the use of effective contraception while on treatment period.
10. Patients must be able to understand and be willing to sign a written informed consent document.
11. Patients must be able to comply with the study protocol.

Exclusion Criteria:

1. Diagnosed as nasopharyngeal cancer.
2. Body mass index (BMI) < 18.5.
3. Significant history of cardiac disease (i.e. uncontrolled hypertension, unstable angina, congestive heart failure, or uncontrolled arrhythmias, etc.).
4. Patients with a history of any other malignancy (except squamous or basal cell skin cancer or cervical carcinoma in situ) are ineligible, unless the patient has been continuously disease-free for at least 5 years.
5. Previously received chemotherapy, radiation therapy, or immunotherapy for head and neck cancer.
6. Dysphagia patients who do not consent to nasogastric (NG), orogastric (OG), or percutaneous endoscopic gastrostomy (PEG) feeding.
7. History or clinical evidence of any hyperthyroidism, cirrhosis, hepatic failure, human immunodeficiency virus (HIV) infection, renal failure (as determined by a serum creatinine > 250 µmol/L or > 2.83 mg/dL at screening), active tuberculosis (as confirmed by sputum or other microbiological methods within the last five years), or active hepatitis B/C.
8. Any other clinical disorders or unsuitable conditions that render the patient ineligible for this study, as determined by the principal investigator(s).
9. Treatment with any investigational product or health supplement within 28 days prior to enrollment.
10. Pregnant or breastfeeding women.
11. Non-compliance with the requirement for contraception or other aspects of the study protocol.
12. Inability to understand and provide informed consent regarding participation in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-01-23 (Estimated)

PRIMARY OUTCOMES:
To evaluate disease-free survival (DFS) of patients treated with a combination of fucoidan, chemotherapy, and radiation therapy | From date of randomization and assessed up to 96 weeks
  To evaluate disease-free survival (DFS) of patients treated with a combination of fucoidan, chemotherapy, and radiation therapy

SECONDARY OUTCOMES:
To evaluate pain in patients treated with a combination of fucoidan, chemotherapy, and radiation therapy | From date of randomization to the end of treatment period, up to 24 weeks
  To evaluate pain in patients treated with a combination of fucoidan, chemotherapy, and radiation therapy by a numerical rating scale (NRS: 0-10)
To evaluate the disease control rate (DCR) of patients treated with a combination of fucoidan, chemotherapy, and radiation therapy | From date of randomization and assessed up to 96 weeks
  To evaluate the disease control rate (DCR) of patients treated with a combination of fucoidan, chemotherapy, and radiation therapy

OTHER OUTCOMES:
To evaluate the safety of fucoidan, as defined by the incidence of treatment-emergent adverse events (TEAEs) | From date of randomization to the end of treatment period, up to 24 weeks
  To evaluate the safety of fucoidan, as defined by the incidence of treatment-emergent adverse events (TEAEs)
To evaluate the quality of life (QoL) of patients treated with a combination of fucoidan, chemotherapy, and radiation therapy by using questionnaire: EQ5D | From date of randomization to the end of treatment period, up to 24 weeks
  To evaluate the quality of life (QoL) of patients treated with a combination of fucoidan, chemotherapy, and radiation therapy by using questionnaire: EuroQol five dimensions questionnaire (EQ5D)
To evaluate the quality of life (QoL) of patients treated with a combination of fucoidan, chemotherapy, and radiation therapy by using questionnaire: EORTC QLQ-H&N35 | From date of randomization to the end of treatment period, up to 24 weeks
  To evaluate the quality of life (QoL) of patients treated with a combination of fucoidan, chemotherapy, and radiation therapy by using questionnaire: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module 35 (H&N 35)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jen Lou, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei County, Taiwan